CLINICAL TRIAL: NCT02528305
Title: A Pilot Project to Assess the Effect of High-intensity Interval Training in Patients With Non-alcoholic Fatty Liver Disease/Steatohepatitis
Brief Title: The Effect of HIT in Patients With Non-alcoholic Fatty Liver Disease/Steatohepatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Abertay University (Other)
Responsible Party: Principal Investigator, Niels Vollaard, Lecturer in Human and Applied Physiology, University of Bath
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015CM
Record Dates: First submitted 2015-08-10; First posted 2015-08-19 (Estimated); Results first posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Non-alcoholic Steatohepatitis; Non-alcoholic Fatty Liver Disease
Keywords: High-intensity Interval Training
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — High-Intensity Interval Training; Exercise

STUDY DESIGN:
Masking Description: No Masking, this was not possible with this study design.
Oversight: Data Monitoring Committee: No

ARMS (1):
- High-intensity Interval Training (HIT) (Experimental): 6 week control period with no intervention then 6 weeks of twice weekly HIT
  Interventions: Other: High-intensity Interval Training

INTERVENTIONS:
Other: High-intensity Interval Training — 2 minute warm-up at 50rpm, then increase to 100rpm. Weight added to bike (7% body weight for men 6% body weight for women). Continue effort for 6 seconds, then passive rest for at least 1 minute. Total 5 sprints in sessions 1-3, 6 sprints in session4, 7 sprints in sessions 5&6, 8 sprints in sessions 7&8, 9 sprints in sessions 9&10 and 10 sprints in sessions 11&12.
  Other Names: Exercise

SUMMARY:
This pilot study aims to investigate whether 6 weeks of twice weekly High-intensity Interval Training (HIT) results in improvements in disease-specific measures, feelings of general well-being, physical fitness and cognitive function in patients with non-alcoholic fatty liver disease or non-alcoholic steatohepatitis.

DETAILED DESCRIPTION:
The study aims to recruit up to 12 patients diagnosed with non-alcoholic fatty liver disease (NAFLD) or non-alcoholic steatohepatitis (NASH) from the liver clinics at Ninewells Hospital, Dundee. Suitable patients who give informed consent will be assessed at baseline, again after 6 weeks of no intervention to act as a control period, and thirdly after 6 weeks of twice-weekly high-intensity interval training (HIT).

Assessments will be performed with the patient fasted overnight, and will involve body composition measurements, blood pressure, a venous blood sample for circulating triglycerides, fasting glucose, insulin, liver enzymes alanine aminotransferase (ALT) and aspartate aminotransferase (AST), and platelets. An oral glucose tolerance test will be performed using fingerprick capillary samples. Cognitive function tests for episodic memory, executive function and semantic memory will be performed and a questionnaire (SF-36) will be used to assess general well-being. Physical fitness will be assessed through a 12-minute walk test on a treadmill, which will allow estimation of maximal oxygen uptake capacity (VO2 max), and a "get up and go" test will be used to assess physical function.

The exercise intervention will involve a 2 minute warm-up, cycling at 50 rpm before the participants will be asked to cycle at 100rpm and a weight will be added (7% body weight for men and 6% body weight for women) as resistance. The sprint will last 6 seconds and the participant will be asked to rest for at least 1 minute. This will be repeated for a total of 5 sprints in sessions 1-3, 6 sprints in session 4, 7 sprints in sessions 5&6, 8 sprints in sessions 7&8, 9 sprints in sessions 9&10 and 10 sprints in sessions 11&12. Exercise heart rate will be monitored and recorded.

At least 3 days after the last HIT session the pre-intervention testing assessment will be repeated for a third time.

Changes in measured variables will be analysed via repeated measures analysis of variance (ANOVA) with post-hoc testing of all variables.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of non-alcoholic fatty liver disease or non-alcoholic steatohepatitis
* attending a specialist liver clinic at Ninewells Hospital, Dundee

Exclusion Criteria:

* unstable cardiovascular disease
* uncontrolled arrhythmias
* structural cardiac abnormalities
* uncontrolled diabetes
* other uncontrolled metabolic abnormalities
* severe orthopaedic condition that would prohibit exercise
* severe pulmonary condition that would prohibit exercise
* any other poorly controlled medical condition.
* resting systolic blood pressure above 160 mm Hg
* resting diastolic blood pressure above 90 mm Hg
* symptomatic postural drop in blood pressure greater than 20 mm Hg

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niels BJ Vollaard, PhD, Principal Investigator — University of Bath
Locations (2):
- United Kingdom (2):
  - Abertay University, Dundee
  - Ninewells Hospital, Dundee

IPD SHARING:
Plan to Share IPD: No
There is no reason to share the IPD.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-intensity Interval Training (HIT)
Started | 12
End of Control Period Assessment | 11
End of Intervention Period Assessment | 9
Completed | 9
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | High-intensity Interval Training (HIT)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
height [Mean (Standard Deviation); unit: metres] | 1.71 (0.09)
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (3.8)
diagnosis [Number; unit: participants]
  Non-alcoholic Fatty Liver Disease (NAFLD) | 7
  Non-alcoholic Steatohepatitis (NASH) | 5

OUTCOME MEASURES:

1. Primary Outcome: Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: calculation of insulin resistance via formula: fasting insulin (mIU/L) x fasting glucose (mg/dL)/405 normal insulin resistance -HOMA score <3 moderate insulin resistance -HOMA score 3-5 severe insulin resistance -HOMA score >5 Assessed at baseline, after 6 week control period and within 1 week of completing 6 weeks HIT
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Baseline Assessment: on entry to trial
- After 6 Week Control Period: repeat assessment after 6 weeks of no intervention
- After HIT Assessment: final assessment within 1 week of completing 6 weeks of HIT
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
units on a scale | 6.9 (4.7) | 9.6 (10.5) | 7.0 (4.3)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.474, ANOVA

2. Primary Outcome: Oral Glucose Tolerance Test
Description: measurement of capillary samples for glucose at time 0, followed by every 20 minutes for 2 hours following ingestion of 75g glucose. Results graphed against time, then area under the curve calculated for each of the 3 assessments.
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: mmol/L*min
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
mmol/L*min | 981 (136) | 1030 (182) | 1010 (247)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.174, ANOVA

3. Primary Outcome: AST: ALT Ratio
Description: ratio of liver enzymes aspartate aminotransferase (AST) to alanine aminotransferase (ALT).
  used as a diagnostic aid e.g. AST:ALT of more than 2:1 is characteristic of alcoholic liver disease whereas fatty steatosis and many other causes of liver disease, ratio is less than or equal to 1.
  Ratio may rise as fibrosis and cirrhosis develop in viral hepatitis.
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
ratio | 0.5 (0.2) | 0.5 (0.2) | 0.5 (0.2)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.303, ANOVA

4. Primary Outcome: FIB-4
Description: calculated from AST, ALT, platelets and participant's age and used to estimate amount of fibrosis in liver.
  Fib-4 score of <1.45 has negative predictive value of 90% for advanced fibrosis.
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: Fibrosis Score
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
Fibrosis Score | 0.68 (0.18) | 0.60 (0.19) | 0.60 (0.18)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority; p = 0.023, ANOVA

5. Primary Outcome: Body Fat Mass Estimated Via Bioimpedance
Description: total body fat and trunk fat estimated via bioimpedance measured after overnight fast, expressed as percentage
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: percentage body fat
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
percentage body fat
  total fat | 29.7 (8.2) | 29.5 (8.3) | 28.3 (7.1)
  trunk fat | 26.6 (6.0) | 29.1 (5.4) | 28.6 (5.7)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.092, ANOVA; For the analysis of Total body fat
Statistical Analysis 2: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.101, ANOVA; For the analysis of Trunk fat

6. Primary Outcome: Blood Pressure
Description: taken with participant supine, measured on left arm
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
mmHg
  systolic blood pressure | 139 (18) | 142 (13) | 136 (19)
  diastolic blood pressure | 85 (13) | 87 (10) | 78 (8)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.771, ANOVA; For the analysis of systolic blood pressure
Statistical Analysis 2: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.028, ANOVA; For the analysis of diastolic blood pressure

7. Primary Outcome: General Well-being as Assessed by SF-36 Questionnaire
Description: Assessment of: physical functioning, social functioning, mental health, pain, change in health, physical role limitation, mental role limitation, energy and vitality, health perception over preceding 4 weeks (other than change in health, which is a comparison to health the preceding year), expressed as a transformed score range 0-100, with a higher score indicating better function/freedom from pain etc
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
units on a scale
  Physical Function | 79 (25) | 85 (22) | 92 (16)
  Social Function | 78 (31) | 82 (27) | 83 (27)
  Mental Health | 71 (17) | 69 (20) | 77 (20)
  Pain | 78 (13) | 72 (28) | 88 (16)
  Change in Health | 50 (18) | 53 (15) | 67 (18)
  Physical Role Limitation | 79 (27) | 79 (31) | 90 (22)
  Mental Role Limitation | 76 (24) | 76 (34) | 81 (30)
  Energy/Vitality | 58 (18) | 56 (20) | 64 (21)
  Health Perception | 58 (19) | 60 (17) | 61 (17)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.099, ANOVA; For the analysis of Physical Function
Statistical Analysis 2: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.566, ANOVA; For the analysis of Social Function
Statistical Analysis 3: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.246, ANOVA; For the analysis of Mental Health
Statistical Analysis 4: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.145, ANOVA; For the analysis of Pain
Statistical Analysis 5: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.085, ANOVA; For the analysis of Change in Health
Statistical Analysis 6: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.114, ANOVA; For the analysis of Physical Role Limitation
Statistical Analysis 7: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.841, ANOVA; For the analysis of Mental Role Limitation
Statistical Analysis 8: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.366, ANOVA; For the analysis of Energy/Vitality
Statistical Analysis 9: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.745, ANOVA; For the analysis of Health Perception

8. Primary Outcome: Short-term Memory Recall
Description: testing of verbal word presentation-immediate recall of 10 words (60 seconds for recall) Maximum =10, minimum =0
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
words | 6 (2) | 7 (1) | 6 (2)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.310, ANOVA

9. Primary Outcome: Estimated VO2 Max
Description: VO2 max estimated via submaximal exercise test-submaximal treadmill walking test Calculated via formula: VO2max= 15.1+21.8 x speed (miles per hour) - 0.327 x heart rate (beats per minute) - 0.263 x speed x age (years) + 0.00504 x heart rate x age + 5.98 x gender (0=female, 1=male)
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: millilitres/kilogram/minute
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
millilitres/kilogram/minute | 34.9 (6.5) | 37.6 (7.2) | 38.5 (7.2)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p < 0.001, ANOVA

10. Primary Outcome: Physical Function-"Get up and go" Test
Description: participant will be timed standing up from chair unaided,walking 30m, turning round and returning to a seated position on the chair, the average time of 3 attempts will be recorded.
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
seconds | 6.61 (0.77) | 6.23 (0.59) | 5.87 (0.63)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.005, ANOVA

11. Primary Outcome: Ankle Brachial Pressure Index (ABPI)
Description: ratio of blood pressure in left arm and right ankle
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: ABPI
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
ABPI | 1.15 (0.16) | 1.08 (0.18) | 1.13 (0.27)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.793, ANOVA

12. Primary Outcome: Long-term Memory Recall
Description: testing of verbal word presentation-delayed recall of 10 words 10 minutes after words initially presented (within 60 seconds).
  Maximum= 10 words, minimum = no words
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
words | 4 (1) | 5 (2) | 5 (2)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.513, ANOVA

13. Primary Outcome: Executive Function (Verbal Fluency Test)
Description: written verbal fluency test: participant asked to write down as many English words as possible within 60 seconds, starting with a particular letter of the alphabet, excluding proper nouns or plurals.
  Baseline assessment-letter A Post Control assessment -letter S After HIT assessment -letter F
Time Frame: Baseline, Follow up at 6 Weeks and following HIT intervention at 12 Weeks
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Baseline Assessment | After 6 Week Control Period | After HIT Assessment
Number analyzed (Participants) | 9 | 9 | 9
words | 8 (4) | 12 (4) | 11 (3)
Statistical Analysis 1: Comparison: Baseline Assessment vs After 6 Week Control Period vs After HIT Assessment; Test type: Superiority or Other; p = 0.009, ANOVA

ADVERSE EVENTS:
Arm/Group | High-intensity Interval Training (HIT)
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-intensity Interval Training (HIT) (N=12)
Myocardial Infarction (Cardiac disorders) | 1 (1) — occurred at home during 6 week period of HIT intervention. Cardiologist concluded HIT had not contributed to his infarction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes